CLINICAL TRIAL: NCT07073469
Title: Tenecteplase in ReperfUsion Therapy for Posterior Circulation Stroke With Extended Time Window: the TRUST Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Min Lou, Dr., Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRUST
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Stroke Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Tenecteplase with standard therapy (Experimental): Patients will receive standard dose intravenous tenecteplase (0.25 mg per kilogram, with a maximum dose of 25 mg)
  Interventions: Drug: Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg)
- Standard therapy (Active Comparator): Standard therapy
  Interventions: Other: Standard medical treatment

INTERVENTIONS:
Drug: Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg) — Tenecteplase (TNK) (0.25 mg/kg, to maximum of 25mg)
  Arms: Experimental: Tenecteplase with standard therapy
Other: Standard medical treatment — Standard medical treatment according to local guidelines
  Arms: Standard therapy

SUMMARY:
The primary hypothesis being tested in this trial is that ischemic stroke patients in posterior circulation at 4.5 - 24 hours post onset of stroke will have improved clinical outcomes when given intravenous TNK compared to standard care.

DETAILED DESCRIPTION:
Posterior circulation stroke accounts for 20-25% of all ischemic strokes, with an annual adjusted incidence of 18 per 100,000 person-years. Compared with anterior circulation stroke, posterior circulation stroke is less studied and has poor neurological outcomes, which requires attention. Intravenous thrombolytic therapy has greatly improved the rate of recanalization and reperfusion in patients with acute ischemic stroke, increased the proportion of patients with good prognosis, and reduced mortality. Guidelines recommend intravenous thrombolysis within 4.5 hours of onset or awakening in patients with ischemic stroke. However, the proportion of posterior circulation stroke is low or unreported in most randomized controlled trials, such as 5% of patients in the NINDS study, so it may be inappropriate to apply the results of these trials directly to patients with posterior circulation ischemic stroke.

Multiple studies have also shown a lower risk of post-circulation bleeding complications compared to pre-circulation stroke. A meta-analysis of patients with posterior circulation ischemic stroke (11.9% of posterior circulation stroke) showed that posterior circulation stroke had a lower risk of intracranial hemorrhage due to intravenous thrombolysis, half the risk of anterior circulation stroke, and a higher 3-month good functional outcome. The lower risk of hemorrhagic transformation in posterior circulation stroke is due to the greater tolerance of the posterior circulation area to ischemic injury, possibly due to a greater proportion of white matter and arterial collaterals, especially in the brainstem. In addition, the smaller infarct size of posterior circulation stroke compared with anterior circulation stroke also reduced the risk of bleeding in these patients.

Our previous EXPECTs trial have proved the effectiveness and safety of intravenous alteplase in patients with posterior circulation stroke within 4.5-24 hours of onset. However, the effectiveness of tenecteplase (TNK) has not been studied in this subgroup of patients. Therefore, the purpose of this study was to investigate whether patients with posterior circulation stroke with onset or discovery time of 4.5-24 hours could benefit from intravenous TNK in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with clinical signs of acute ischemic stroke between 4.5 and 24 hours from stroke onset, or wake-up stroke and unwitnessed stroke (if the midpoint of the last known well time is within 4.5 to 24 hours)
2. Patients aged > 18 years (or as per local requirements)
3. NIHSS ≥ 4
4. Patients with a posterior circulation ASPECT score (PC-ASPECTS) ≥ 7. If MRI is performed first and the PC-ASPECTS on diffusion-weighted imaging (DWI) is ≥ 7, a non-contrast head CT is not required. If PCASPECTS on DWI is < 7, the subsequent non-contrast CT must show a PC-ASPECTS ≥ 7 for inclusion
5. Posterior circulation stroke confirmation criteria: If MRI is performed, infarction confirmed by DWI is sufficient. If CT is performed, the non-contrast CT scan must not refute posterior circulation stroke, and clinical signs and symptoms must support the diagnosis, as confirmed by experienced clinicians. If clinical symptoms are atypical, CTA showing symptomatic stenosis or occlusion of large posterior circulation vessels, or CT perfusion showing symptomatic hypoperfusion, can provide additional evidence, though advanced imaging is not mandatory
6. Pre-stroke mRS score < 2
7. Informed consent has been obtained from the patient, a family member, or a legally responsible person, depending on local ethics requirements

Exclusion Criteria:

1. Contraindications for tenecteplase:

   * Allergy to tenecteplase
   * Rapidly improving symptoms at the discretion of the investigator
   * The presence of epileptic seizures, hemiplegia after seizures (Todd's palsy), or other neurological/mental illnesses that prevent cooperation or willingness to participate
   * Persistent blood pressure elevation (systolic ≥180 mmHg or diastolic ≥100 mmHg) despite treatment
   * Blood glucose levels outside the acceptable range (<2.8 mmol/L or >22.2 mmol/L), with point-of-care glucose testing considered valid
   * High risk of bleeding due to active internal bleeding, major surgery, trauma, gastrointestinal, or urinary tract hemorrhage within the previous 21 days, or arterial puncture at a non-compressible site within the previous 7 days
   * Known impairments in coagulation due to comorbid disease or anticoagulant use, including an INR >1.7 or prothrombin time >15 seconds for those on warfarin, recent use of direct thrombin inhibitors or direct factor Xa inhibitors without reversal capability, or full-dose heparin/heparinoid within the last 24 hours with an aPTT above normal limits
   * Known defect in platelet function or a platelet count below 100,000/mm³
   * History of ischemic stroke, myocardial infarction, intracranial hemorrhage, severe traumatic brain injury, or intraspinal operation within the previous 3 months, or known intracranial neoplasm, arteriovenous malformation, or giant aneurysm
   * Acute or past intracerebral hemorrhage identified by CT or MRI
2. Infarction of the anterior circulation confirmed by MRI, or vascular examination indicating occlusion of large anterior circulation vessels, or perfusion imaging showing hypoperfusion changes in the anterior circulation area
3. Pregnancy, nursing, or unwillingness to use effective contraceptive measures during the trial period
4. Likelihood of non-adherence to the trial protocol or follow-up
5. Any condition that, in the judgment of the investigator, could impose hazards if study therapy is initiated or affect patient participation in the study
6. Participation in other interventional clinical trials within the previous 3 months
7. A life expectancy of less than three months
8. The judgment is left to the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Ordinal distribution of modified Rankin Scale (mRS) score at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome

SECONDARY OUTCOMES:
Excellent recovery assessed by the ratio of modified Rankin Scale (mRS) score of 0-1 (%) at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
Independent recovery assessed by ratio of modified Rankin Scale (mRS) score of 0-2 (%) at 90 ± 7 days | 90 ± 7 days
  mRS: minimum value = 0, maximum value = 6, and lower scores mean a better outcome
Major neurologic improvement (%) at 24 hours defined as an improvement on National Institutes of Health Stroke Scale (NIHSS) score ≥ 8 points compared with the initial deficit or a score ≤ 1 | 24 hours
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
Major neurologic improvement (%) at 7 days defined as an improvement on National Institutes of Health Stroke Scale (NIHSS) score ≥ 8 points compared with the initial deficit or a score ≤ 1 | 7 days
  NIHSS: minimum value = 0, maximum value = 42, and higher scores mean severer symptoms
Symptomatic intracerebral hemorrhage (sICH) within 36 hours after randomization | within 36 hours
  sICH as defined by The European Cooperative Acute Stroke Study III criteria [ECASSIII]
Parenchymal hematoma (PH) (%) within 36 hours after randomization | within 36 hours
  PH as defined by the European Cooperative Acute Stroke Study [ECASS] criteria
Any intracerebral hemorrhage (ICH) within 36 hours after randomization | within 36 hours
Mortality (%) within 90 days | 90 days
  Mortality refers to rate of death from any cause